CLINICAL TRIAL: NCT00908076
Title: Randomized Double-Blind Placebo-Controlled Trial of Lubiprostone in the Treatment of Constipation Associated With Parkinson's Disease
Brief Title: Amitiza in Constipation Associated With PD (Parkinson's Disease)
Acronym: AMITIZA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of South Florida (Other)
Responsible Party: Principal Investigator, Joseph Jankovic, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-21192; NCT00849784 (obsolete NCT alias)
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Results first posted 2016-08-26 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Parkinson's Disease
Keywords: constipation; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Constipation | interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- amitiza (Active Comparator): Amitiza
  Interventions: Drug: LUBIPROSTONE
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: LUBIPROSTONE

INTERVENTIONS:
Drug: LUBIPROSTONE — Subjects will be randomized into placebo and study groups. Half of the study group (N=39) will be given lubiprostone (24 mcg) twice daily; the other half will receive matching placebo twice daily.

SUMMARY:
The purpose of this study is to determine if Amitiza (lubiprostone), a drug proven to be safe and effective for chronic constipation, will also improve constipation symptoms in Parkinson's Disease patients. We will also evaluate the impact of the drug on changes in bowel movement consistency, quality of life and motor symptoms.

DETAILED DESCRIPTION:
Parkinson's disease (PD) affects about one million people in the United States. It is a common neurological condition that is clinically defined by rigidity (muscle stiffness), bradykinesia (slowness of movement) and tremor. Parkinson's Disease , however, reveals numerous non-motor symptoms that have been underemphasized. Problematic symptoms include varying degrees of dementia, psychosis, diminished assertiveness and confidence, general fatigue, excessive daytime sleepiness, problems with blood pressure, sweating, and bladder, and a common yet difficult to define sense of "not feeling well".

A commonly missed symptom in Parkinson's patients is constipation. Constipation can be difficult to treat with current medications available and many are ineffective. Levodopa and dopamine agonists drugs are useful for motor symptoms in Parkinson's Disease but have no effect on constipation. Laxatives and enemas provide limited relief with bothersome side effects. Even fewer drugs have been studied targeting the constipation problem specifically in the Parkinson's Disease population. Lubiprostone (AMITIZA) is a new medication that has been studied in the general population for the treatment of chronic constipation. It has been shown to be a safe and effective medication with few side effects. Lubiprostone has not yet been studied in the Parkinson's Disease population. We hope to show that this medication can be safe and effective for constipation in PD patients as well.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects must be diagnosed with PD according to conventional criteria.
* 2. Subjects must report having constipation and fulfill Rome III criteria19 for chronic constipation: at least 3 months, in the last 6 months with two or more of the following: i. Less than 3 SBM's per week ii. Straining with defecation more than 25% of the time iii. Lumpy or hard stools with defecation more than 25% of the time iv. Sensation of incomplete evacuation with defecation more than 25% of the time v. Sensation of anorectal obstruction or blockage with defecation more than 25% of the time vi. Use of manual maneuvers to facilitate defecation more than 25% of the time
* 3. Patients will be encouraged to use only lubiprostone for constipation. If they use any other agents they will need to record this use in their diary; any BM that occurs within 24 hours of the other agent used will be recorded, but not be counted as a SBM.
* 4. Patients or patients' caretaker(s)/ legal guardian must be able to read, understand, and accurately record data into the diary to guarantee full participation in the study.
* 5. Patients over the age of 50 must have had a colonoscopy or sigmoidoscopy within 5 years.
* 6. Patients or patient's caretaker(s)/legal guardian must be willing and able to provide informed consent before beginning the study.

Exclusion Criteria:

* Evidence of structural abnormality of the gastrointestinal tract or diseases/conditions that affect bowel transit including gastric, small bowel or colonic resection (appendectomy, cholecystectomy, benign polypectomy are allowed); history of colon cancer, history of inflammatory bowel disease (Crohn's disease or ulcerative colitis); insulin-dependent diabetes mellitus, history of Hirschsprung's disease, progressive systemic sclerosis (scleroderma), anorexia nervosa; other diseases or conditions that in the opinion of the investigator significantly affect bowel transit. Subjects with constipation secondary to any other documented cause.
* Planned use of drugs or agents during pretreatment phase onward that affect gastrointestinal motility and/ or prescription including laxatives including stool softeners (patients experiencing significant constipation may use a laxative as rescue medication if needed); antidiarrheals (in case of significant diarrhea loperamide may be used if needed); antacids containing magnesium or aluminum salts (only calcium containing ones are allowed); anticholinergics, antispasmodic agents (e.g., Librax, Donnatal, dicyclomine); erythromycin and other macrolides; octreotide; ondansetron or other 5-HT3 antagonists; opioids/narcotic analgesics; prokinetics (metoclopramide); serotonin re-uptake inhibitors or tricyclic antidepressants (allowed if constant doses for at least 1 month before treatment); calcium antagonists (allowed if constant doses for at least 1 month before treatment).
* Subjects with any significant cardiovascular, liver, lung, renal, psychiatric or neurological diseases (not including PD).
* Patients with previous allergic reaction or lack of tolerability to lubiprostone.
* Current or recent history (within 12 months) of drug or alcohol abuse.
* Pregnancy or breast feeding.
* Fertile women (defined as those who are not surgically sterile, are not >1 year post-menopausal or who are not currently using or complying with a medically approved method of contraception). Lubiprostone has not been studied in pregnant women and should only be used during a pregnancy if the potential benefits justify the potential risk to the fetus. Women should have a negative pregnancy test before beginning treatment with lubiprostone and need to practice effective contraceptive measures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G Ondo, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - University of South Florida, Tampa, Florida
  - Baylor College of Medicine PDCMDC, Houston, Texas

REFERENCES:
- [Background] Ondo WG, Kenney C, Sullivan K, Davidson A, Hunter C, Jahan I, McCombs A, Miller A, Zesiewicz TA. Placebo-controlled trial of lubiprostone for constipation associated with Parkinson disease. Neurology. 2012 May 22;78(21):1650-4. doi: 10.1212/WNL.0b013e3182574f28. Epub 2012 May 9. PMID 22573627

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amitiza | Placebo
Started | 27 | 27
Completed | 26 | 26
Not Completed | 1 | 1
Not completed — Lack of Efficacy | 1 | 1

BASELINE CHARACTERISTICS:
Population: Patients were included if they had PD using standard criteria, were aged 35 to 85 years, and met the ROME II criteria19 and scored at least 10 on the ROME II constipation assessment. Excluded if they had any other identifiable cause of constipation, use of opioids, anticholinergic agents, or antacids containing magnesium or aluminum salts.
Groups:
- Total: Total of all reporting groups
Arm/Group | Amitiza | Placebo | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (8.1) | 70.1 (12.2) | 68.0 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 20 | 19 | 39
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54
PD duration [Mean (Standard Deviation); unit: years] | 8.9 (6.3) | 9.5 (6.3) | 9.2 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Study
Description: Global impression of change, stool diary, visual analog scale of improvement, UPDRS rating scale and constipation questionnaires. The primary efficacy data will be analyzed using Student's t-test with unequal variances as the difference from baseline in SBM comparing cases and controls, using last observation carried forward for missing data in the intent-to-treat population.
Time Frame: Baseline to end of study
Population: A marked or very marked clinical global improvement.
  Ondo WG et al. Placebo-controlled trial of lubiprostone for constipation associated with Parkinson disease. Neurology 2012 May 22; 78:1650. - See more at: http://www.jwatch.org/jn201205290000006/2012/05/29/lubiprostone-constipation-parkinson-disease#sthash.ggWrS7Vq.dpuf
Measure: Number; unit: Percentage of participants
Arm/Group | Amitiza | Placebo
Number analyzed (Participants) | 27 | 27
Percentage of participants | 64 | 18.5

ADVERSE EVENTS:
Groups:
- Amitiza; Placebo: LUBIPROSTONE: Subjects will be randomized into placebo and study groups. Half of the study group (N=27) will be given lubiprostone (24 mcg) twice daily; the other half will receive matching placebo twice daily.
Arm/Group | Amitiza | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 3/27 | 1/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amitiza (N=27) | Placebo (N=27)
diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No